CLINICAL TRIAL: NCT02772770
Title: Pediatric ACL: Understanding Treatment Options (PLUTO)
Brief Title: Pediatric ACL: Understanding Treatment Options
Acronym: PLUTO
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Children's Hospital Medical Center, Cincinnati (Other); Rady Children's Hospital, San Diego (Other); Washington University School of Medicine (Other); Children's Healthcare of Atlanta (Other); The Cleveland Clinic (Other); Tennessee Orthopedic Alliance (Other); Hospital for Special Surgery, New York (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Mininder Kocher, Principal Investigator, Boston Children's Hospital
Other Study IDs: IRB-P00017850
Record Dates: First submitted 2016-05-11; First posted 2016-05-16 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Anterior Cruciate Ligament Reconstruction
MeSH Terms: interventions — Braces

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Non Operative: Rehabilitation, Bracing, Activity Restriction
  Interventions: Other: Non-operative treatment group will undergo standardized treatment which will include rehabilitation, bracing and certain activity restrictions
- Operative: Transphyseal
  Interventions: Procedure: Surgical technique: Transphyseal reconstruction
- Operative: Partial Transphyseal
  Interventions: Procedure: Surgical technique: Partial transphyseal reconstruction
- Operative: Physeal sparing by Anderson Technique
  Interventions: Procedure: Surgical technique: Physeal sparing reconstruction by the Anderson method
- Operative: Physeal sparing by Micheli/Kocher Technique
  Interventions: Procedure: Surgical technique: Physeal sparing reconstruction by the Micheli/Kocher method

INTERVENTIONS:
Other: Non-operative treatment group will undergo standardized treatment which will include rehabilitation, bracing and certain activity restrictions — The non-operative treatment group will undergo standardized treatment which will include rehabilitation, bracing and certain activity restrictions.
  Groups: Non Operative: Rehabilitation, Bracing, Activity Restriction
Procedure: Surgical technique: Transphyseal reconstruction — Study physicians will have the option to treat ACL injuries operatively or non-operatively, according to their standard of care. However, once the decision is made to manage the injury operatively or non-operatively, the physician must follow the appropriate standardized treatment protocol developed for the study. The operative treatment protocol will include standardized surgical techniques for transphyseal reconstruction with soft tissue graft and metaphyseal fixation.
  Groups: Operative: Transphyseal
Procedure: Surgical technique: Partial transphyseal reconstruction — Study physicians will have the option to treat ACL injuries operatively or non-operatively, according to their standard of care. However, once the decision is made to manage the injury operatively or non-operatively, the physician must follow the appropriate standardized treatment protocol developed for the study. The operative treatment protocol will include partial transphyseal reconstruction (tibial transphyseal and femoral epiphyseal) with soft tissue graft.
  Groups: Operative: Partial Transphyseal
Procedure: Surgical technique: Physeal sparing reconstruction by the Anderson method — Study physicians will have the option to treat ACL injuries operatively or non-operatively, according to their standard of care. However, once the decision is made to manage the injury operatively or non-operatively, the physician must follow the appropriate standardized treatment protocol developed for the study. The operative treatment protocol will include standardized surgical techniques for physeal sparing epiphyseal reconstruction with soft tissue graft (Anderson technique).
  Groups: Operative: Physeal sparing by Anderson Technique
Procedure: Surgical technique: Physeal sparing reconstruction by the Micheli/Kocher method — Study physicians will have the option to treat ACL injuries operatively or non-operatively, according to their standard of care. However, once the decision is made to manage the injury operatively or non-operatively, the physician must follow the appropriate standardized treatment protocol developed for the study. The operative treatment protocol will include physeal-sparing with Iliotibial band combined extra-articular and intra-articular reconstructions (Micheli/Kocher Technique).
  Groups: Operative: Physeal sparing by Micheli/Kocher Technique

SUMMARY:
Pediatric ACL: Understanding Treatment Outcomes (PLUTO) is a multi-center, prospective cohort study. Specific aims of PLUTO are to evaluate the safety and comparative effectiveness of non-operative treatment, as well as four operative treatments including (1) transphyseal ACL reconstruction (2) partial transphyseal ACL reconstruction, (3) physeal-sparing epiphyseal ACL reconstruction using the Anderson technique, and (4) physeal-sparing ACL reconstruction using the Micheli/Kocher technique in prepubescent and pubescent skeletally immature patients.

DETAILED DESCRIPTION:
Anterior Cruciate Ligament (ACL) injuries are being seen with increased frequency in pediatric and adolescent patients. The management of these injuries is controversial and includes nonoperative treatment and operative treatment with various surgical techniques. Pediatric ACL: Understanding Treatment Outcomes (PLUTO) is a multi-center, prospective cohort study. Specific aims of PLUTO are to evaluate the safety and comparative effectiveness of non-operative treatment, as well as four operative treatments including (1) transphyseal ACL reconstruction (2) partial transphyseal ACL reconstruction, (3) physeal-sparing epiphyseal ACL reconstruction using the Anderson technique, and (4) physeal-sparing ACL reconstruction using the Micheli/Kocher technique in prepubescent and pubescent skeletally immature patients. Accrual will take place over eight years at 9 pediatric sports medicine centers. Post-treatment outcome assessment will be performed at 6-9 months, 1 year, and 2, 5, and 10 years after treatment , including functional outcome, activity level, health-related quality of life, graft survivorship, knee stability, knee motion, and growth disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of complete intrasubstance ACL tear
* Skeletally Immature (by knee radiographs)

Exclusion Criteria:

* Prior ACL surgery on the ipsilateral knee
* Congenital ACL deficiency
* Multiple ligament reconstruction required
* Other significant comorbidities including syndromic conditions, neuromuscular disorders or developmental delay
* If scheduling of the ACL surgery is impacted by the skeletal maturity of the patient
* Simultaneous bilateral ACL tears

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The pool of patients for this study will be patients seen in outpatient and sports medicine clinics at each clinical center. The minimum accrual target for this study is 360 surgical patients and 45 non-operative patients
Sampling Method: Non-Probability Sample
Enrollment: 765 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Knee functional outcome at 2 years post-ACL reconstruction (Pedi-IKDC) | 2 years
  To compare outcomes associated with four surgical techniques performed to treat complete intrasubstance ACL tears in pre- and early pubescent children: (1) transphyseal ACL reconstruction (2) partial transphyseal ACL reconstruction, (3) physeal-sparing epiphyseal ACL reconstruction using the Anderson technique, and (4) physeal-sparing ACL reconstruction using the Micheli/Kocher technique.

SECONDARY OUTCOMES:
Health-related quality of life (Pediatric Quality of Life Inventory (PedsQL) | 2 years
  To compare outcomes associated with four surgical techniques performed to treat complete intrasubstance ACL tears in pre- and early pubescent children: (1) transphyseal ACL reconstruction (2) partial transphyseal ACL reconstruction, (3) physeal-sparing epiphyseal ACL reconstruction using the Anderson technique, and (4) physeal-sparing ACL reconstruction using the Micheli/Kocher technique.
Graft failure (MRI, Lachman, Pivot-Shift) | 2 years
  To compare outcomes associated with four surgical techniques performed to treat complete intrasubstance ACL tears in pre- and early pubescent children: (1) transphyseal ACL reconstruction (2) partial transphyseal ACL reconstruction, (3) physeal-sparing epiphyseal ACL reconstruction using the Anderson technique, and (4) physeal-sparing ACL reconstruction using the Micheli/Kocher technique.
Activity level (P-FABS and Physical Activity Questionnaire) | 2 years
  To compare outcomes associated with four surgical techniques performed to treat complete intrasubstance ACL tears in pre- and early pubescent children: (1) transphyseal ACL reconstruction (2) partial transphyseal ACL reconstruction, (3) physeal-sparing epiphyseal ACL reconstruction using the Anderson technique, and (4) physeal-sparing ACL reconstruction using the Micheli/Kocher technique.
Growth disturbance (angular deformity, leg length discrepancy per clinical exam and radiographs) | 2 years
  To compare outcomes associated with four surgical techniques performed to treat complete intrasubstance ACL tears in pre- and early pubescent children: (1) transphyseal ACL reconstruction (2) partial transphyseal ACL reconstruction, (3) physeal-sparing epiphyseal ACL reconstruction using the Anderson technique, and (4) physeal-sparing ACL reconstruction using the Micheli/Kocher technique.

OTHER OUTCOMES:
Re-injury or instability requiring ACL reconstruction | 2 years
  To establish outcomes associated with non-operative treatment (rehabilitation, bracing and activity restriction) used to manage complete intrasubstance ACL tears in pre- and early pubescent children.
Knee function (Pedi-IKDC) | 2 years
  To establish outcomes associated with non-operative treatment (rehabilitation, bracing and activity restriction) used to manage complete intrasubstance ACL tears in pre- and early pubescent children.
Health-related quality of life (PedsQL) | 2 years
  To establish outcomes associated with non-operative treatment (rehabilitation, bracing and activity restriction) used to manage complete intrasubstance ACL tears in pre- and early pubescent children.
Activity level ( P-FABS and Physical Activity Questionnaire) | 2 years
  To establish outcomes associated with non-operative treatment (rehabilitation, bracing and activity restriction) used to manage complete intrasubstance ACL tears in pre- and early pubescent children.
Subsequent meniscal or chondral injury (MRI) | 2 years
  To establish outcomes associated with non-operative treatment (rehabilitation, bracing and activity restriction) used to manage complete intrasubstance ACL tears in pre- and early pubescent children.

CONTACTS AND LOCATIONS:
Overall Officials: Mininder S Kocher, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (10):
- United States (10):
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University at St. Louis, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No